CLINICAL TRIAL: NCT03164356
Title: Portable Bioimpedance Monitoring: Testing a New Diagnostic Interface
Brief Title: Bioimpedance as a Diagnostic Tool for Assessing the Need for Socket Modification in Transtibial Amputees
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Joan Sanders, Professor, Bioengineering, University of Washington
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Diagnostic
Other Study IDs: STUDY00000969
Record Dates: First submitted 2017-03-16; First posted 2017-05-23 (Actual); Results first posted 2022-04-22 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-04

CONDITIONS: Transtibial Amputee
Keywords: Limb Fluid Volume Management; Prosthetic Socket Modification

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Arm 1 (No Intervention): In Arm 1, bioimpedance measurements are taken by research staff. The participants also wear an ActiGraph monitor for at least one week prior to their prosthetist preforming modifications to their socket.
- Arm 2 - Experimental (Experimental): Conclusions drawn from data gathered in Arm 1 will be given to the participant's prosthetist, along with their bioimpedance data from Arm 2, to inform the practitioner's decision on when a modification to the socket is warranted. The results will be compared to those of Arm 3.
  Interventions: Device: Bioimpedance monitor
- Arm 3 - Control (No Intervention): Bioimpedance data will be collected from participants in Arm 3 in parallel with those in Arm 2. However, no data will be provided to the participant's prosthetist.

INTERVENTIONS:
Device: Bioimpedance monitor — Participant in aim 1 will be monitored using the bioimpedance monitor. Data obtained from the arm 1 cohort will be used to inform socket modifications made for arm 2 cohort.
  Arms: Arm 2 - Experimental

SUMMARY:
The purpose of the proposed study is to conduct research on individuals with lower limb amputation, evaluating if residual limb fluid volume data collected using a novel non-invasive device is beneficial towards prosthetic prescription, fit, and comfort as determined by amputee test subjects and practitioners (prosthetists). Participants' residual limb fluid volume will be monitored through bioimpedance analysis both before and after a practitioner-issued modification to the prosthesis as an observational cohort study and then as a blinded randomized control trial in which the data may or may not be shared with the practitioner before the modification is made to the prosthesis.

ELIGIBILITY:
Inclusion Criteria:

* Transtibial amputees, unilateral or bilateral
* Amputation at least 18 months prior
* Walking activity of at least 7 hours per week
* Medicare functional classification level of 2 or higher
* Residual limb length of at least 9 centimeters
* Detrimental impacts to socket fit caused by residual limb volume fluctuations
* Indication for augmented suspension, socket modification/change, sock application removal or activity modification

Exclusion Criteria:

* Incidence of skin breakdown
* Inability to ambulate continuously on a level walkway

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2016-11-09 (Actual); Primary Completion 2020-09-14 (Actual); Study Completion 2020-12-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joan E Sanders, PhD, Principal Investigator — University of Washington
Locations (1):
- University of Washington Bioengineering, Seattle, Washington, United States

REFERENCES:
- [Background] Sanders JE, Severance MR, Allyn KJ. Computer-socket manufacturing error: how much before it is clinically apparent? J Rehabil Res Dev. 2012;49(4):567-82. doi: 10.1682/jrrd.2011.05.0097. PMID 22773260
- [Background] Legro MW, Reiber G, del Aguila M, Ajax MJ, Boone DA, Larsen JA, Smith DG, Sangeorzan B. Issues of importance reported by persons with lower limb amputations and prostheses. J Rehabil Res Dev. 1999 Jul;36(3):155-63. PMID 10659798
- [Background] Kavounoudias A, Tremblay C, Gravel D, Iancu A, Forget R. Bilateral changes in somatosensory sensibility after unilateral below-knee amputation. Arch Phys Med Rehabil. 2005 Apr;86(4):633-40. doi: 10.1016/j.apmr.2004.10.030. PMID 15827911
- [Background] Sanders JE, Cagle JC, Allyn KJ, Harrison DS, Ciol MA. How do walking, standing, and resting influence transtibial amputee residual limb fluid volume? J Rehabil Res Dev. 2014;51(2):201-12. doi: 10.1682/JRRD.2013.04.0085. PMID 24933719
- [Background] Sanders JE, Harrison DS, Allyn KJ, Myers TR, Ciol MA, Tsai EC. How do sock ply changes affect residual-limb fluid volume in people with transtibial amputation? J Rehabil Res Dev. 2012;49(2):241-56. doi: 10.1682/jrrd.2011.02.0022. PMID 22773526
- [Background] Sanders JE, Fatone S. Residual limb volume change: systematic review of measurement and management. J Rehabil Res Dev. 2011;48(8):949-86. doi: 10.1682/jrrd.2010.09.0189. PMID 22068373
- [Background] Van Loan MD, Withers P, Matthie J, Mayclin PL. Use of bioimpedance spectroscopy to determine extracellular fluid, intracellular fluid, total body water, and fat-free mass. Basic Life Sci. 1993;60:67-70. doi: 10.1007/978-1-4899-1268-8_13. No abstract available. PMID 8110166
- [Background] Organ LW, Bradham GB, Gore DT, Lozier SL. Segmental bioelectrical impedance analysis: theory and application of a new technique. J Appl Physiol (1985). 1994 Jul;77(1):98-112. doi: 10.1152/jappl.1994.77.1.98. PMID 7961281
- [Background] Fuller NJ, Hardingham CR, Graves M, Screaton N, Dixon AK, Ward LC, Elia M. Predicting composition of leg sections with anthropometry and bioelectrical impedance analysis, using magnetic resonance imaging as reference. Clin Sci (Lond). 1999 Jun;96(6):647-57. PMID 10334971
- [Background] Salinari S, Bertuzzi A, Mingrone G, Capristo E, Scarfone A, Greco AV, Heymsfield SB. Bioimpedance analysis: a useful technique for assessing appendicular lean soft tissue mass and distribution. J Appl Physiol (1985). 2003 Apr;94(4):1552-6. doi: 10.1152/japplphysiol.00571.2002. PMID 12626475
- [Background] Dittmar M. Reliability and variability of bioimpedance measures in normal adults: effects of age, gender, and body mass. Am J Phys Anthropol. 2003 Dec;122(4):361-70. doi: 10.1002/ajpa.10301. PMID 14614757
- [Background] Andreoli A, Melchiorri G, De Lorenzo A, Caruso I, Sinibaldi Salimei P, Guerrisi M. Bioelectrical impedance measures in different position and vs dual-energy X-ray absorptiometry (DXA). J Sports Med Phys Fitness. 2002 Jun;42(2):186-9. PMID 12032414
- [Background] Donadio C, Consani C, Ardini M, Bernabini G, Caprio F, Grassi G, Lucchesi A, Nerucci B. Estimate of body water compartments and of body composition in maintenance hemodialysis patients: comparison of single and multifrequency bioimpedance analysis. J Ren Nutr. 2005 Jul;15(3):332-44. doi: 10.1016/j.jrn.2005.04.001. PMID 16007563
- [Background] Segal KR, Burastero S, Chun A, Coronel P, Pierson RN Jr, Wang J. Estimation of extracellular and total body water by multiple-frequency bioelectrical-impedance measurement. Am J Clin Nutr. 1991 Jul;54(1):26-9. doi: 10.1093/ajcn/54.1.26. PMID 2058583
- [Background] Wotton MJ, Thomas BJ, Cornish BH, Ward LC. Comparison of whole body and segmental bioimpedance methodologies for estimating total body water. Ann N Y Acad Sci. 2000 May;904:181-6. doi: 10.1111/j.1749-6632.2000.tb06444.x. PMID 10865733
- [Background] Armstrong LE, Kenefick RW, Castellani JW, Riebe D, Kavouras SA, Kuznicki JT, Maresh CM. Bioimpedance spectroscopy technique: intra-, extracellular, and total body water. Med Sci Sports Exerc. 1997 Dec;29(12):1657-63. doi: 10.1097/00005768-199712000-00017. PMID 9432101
- [Background] Siconolfi SF, Gretebeck RJ, Wong WW, Pietrzyk RA, Suire SS. Assessing total body and extracellular water from bioelectrical response spectroscopy. J Appl Physiol (1985). 1997 Feb;82(2):704-10. doi: 10.1152/jappl.1997.82.2.704. PMID 9049756
- [Background] Sanders JE, Rogers EL, Abrahamson DC. Assessment of residual-limb volume change using bioimpedence. J Rehabil Res Dev. 2007;44(4):525-35. doi: 10.1682/jrrd.2006.08.0096. PMID 18247249
- [Background] Sanders JE, Allyn KJ, Harrison DS, Myers TR, Ciol MA, Tsai EC. Preliminary investigation of residual-limb fluid volume changes within one day. J Rehabil Res Dev. 2012;49(10):1467-78. doi: 10.1682/jrrd.2011.12.0236. PMID 23516051
- [Background] Sanders JE, Cagle JC, Harrison DS, Myers TR, Allyn KJ. How does adding and removing liquid from socket bladders affect residual-limb fluid volume? J Rehabil Res Dev. 2013;50(6):845-60. doi: 10.1682/JRRD.2012.06.0121. PMID 24203546
- [Background] Sanders JE, Harrison DS, Cagle JC, Myers TR, Ciol MA, Allyn KJ. Post-doffing residual limb fluid volume change in people with trans-tibial amputation. Prosthet Orthot Int. 2012 Dec;36(4):443-9. doi: 10.1177/0309364612444752. Epub 2012 May 15. PMID 22588848
- [Background] Sanders JE, Hartley TL, Phillips RH, Ciol MA, Hafner BJ, Allyn KJ, Harrison DS. Does temporary socket removal affect residual limb fluid volume of trans-tibial amputees? Prosthet Orthot Int. 2016 Jun;40(3):320-8. doi: 10.1177/0309364614568413. Epub 2015 Feb 20. PMID 25710944
- [Background] Hanspal RS, Fisher K, Nieveen R. Prosthetic socket fit comfort score. Disabil Rehabil. 2003 Nov 18;25(22):1278-80. doi: 10.1080/09638280310001603983. PMID 14617445
- [Background] Legro MW, Reiber GD, Smith DG, del Aguila M, Larsen J, Boone D. Prosthesis evaluation questionnaire for persons with lower limb amputations: assessing prosthesis-related quality of life. Arch Phys Med Rehabil. 1998 Aug;79(8):931-8. doi: 10.1016/s0003-9993(98)90090-9. PMID 9710165
- [Background] Redfield MT, Cagle JC, Hafner BJ, Sanders JE. Classifying prosthetic use via accelerometry in persons with transtibial amputations. J Rehabil Res Dev. 2013;50(9):1201-12. doi: 10.1682/JRRD.2012.12.0233. PMID 24458961
- [Background] Adragao T, Pires A, Branco P, Castro R, Oliveira A, Nogueira C, Bordalo J, Curto JD, Prata MM. Ankle--brachial index, vascular calcifications and mortality in dialysis patients. Nephrol Dial Transplant. 2012 Jan;27(1):318-25. doi: 10.1093/ndt/gfr233. Epub 2011 May 6. PMID 21551082
- [Background] Potier L, Abi Khalil C, Mohammedi K, Roussel R. Use and utility of ankle brachial index in patients with diabetes. Eur J Vasc Endovasc Surg. 2011 Jan;41(1):110-6. doi: 10.1016/j.ejvs.2010.09.020. Epub 2010 Nov 20. PMID 21095144
- [Background] Owings MF, Kozak LJ. Ambulatory and inpatient procedures in the United States, 1996. Vital Health Stat 13. 1998 Nov;(139):1-119. PMID 9866429
- [Background] Pezzin LE, Dillingham TR, Mackenzie EJ, Ephraim P, Rossbach P. Use and satisfaction with prosthetic limb devices and related services. Arch Phys Med Rehabil. 2004 May;85(5):723-9. doi: 10.1016/j.apmr.2003.06.002. PMID 15129395
- [Background] Ziegler-Graham K, MacKenzie EJ, Ephraim PL, Travison TG, Brookmeyer R. Estimating the prevalence of limb loss in the United States: 2005 to 2050. Arch Phys Med Rehabil. 2008 Mar;89(3):422-9. doi: 10.1016/j.apmr.2007.11.005. PMID 18295618
- [Background] Berke GM, Fergason J, Milani JR, Hattingh J, McDowell M, Nguyen V, Reiber GE. Comparison of satisfaction with current prosthetic care in veterans and servicemembers from Vietnam and OIF/OEF conflicts with major traumatic limb loss. J Rehabil Res Dev. 2010;47(4):361-71. doi: 10.1682/jrrd.2009.12.0193. PMID 20803404
- See also: Sandia National Laboratories, Dynamic socket — https://www.sandia.gov/research/dynamic-socket/

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 1 - Pre and Post Modification Observation, No Intervention: In Arm 1, bioimpedance measurements are taken by research staff. The participants also wear an ActiGraph monitor for at least one week prior to their prosthetist preforming modifications to their socket.
- Arm 2 - Treatment Group, Pre and Post Modification: Conclusions drawn from data gathered in Arm 1 will be given to the participant's prosthetist, along with their bioimpedance data from Arm 2, to inform the practitioner's decision on when a modification to the socket is warranted. The results will be compared to those of Arm 3.
- Arm 2 - Control Group, Pre and Post Modification: Bioimpedance data will be collected from participants in Arm 3 in parallel with those in Arm 2. However, no data will be provided to the participant's prosthetist.
- Arm 2 - Prosthetists, Pre and Post Modifications: Participant's in Arm 2 had their prosthetists recruited as well. Prosthetists for participants in both control and treatment groups were surveyed regarding modifications to their patient's socket. Prosthetists for participants in Arm 2 were also given pre-modification bioImpedance data as a supplement to their socket modification process and were surveyed regarding this data as well.
Period: Overall Study
Arm/Group | Arm 1 - Pre and Post Modification Observation, No Intervention | Arm 2 - Treatment Group, Pre and Post Modification | Arm 2 - Control Group, Pre and Post Modification | Arm 2 - Prosthetists, Pre and Post Modifications
Started | 19 | 15 | 17 | 17
Completed | 14 | 10 | 11 | 15
Not Completed | 5 | 5 | 6 | 2
Not completed — Lost to Follow-up | 1 | 1 | 2 | 1
Not completed — Physician Decision | 0 | 0 | 3 | 0
Not completed — Protocol Violation | 2 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0
Not completed — Study timeframe interrupted by Coronavirus disease 2019 (COVID-19) | 1 | 0 | 0 | 1
Not completed — Subject Incarcerated | 0 | 1 | 0 | 0
Not completed — Prosthetist unable to participate | 0 | 2 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Arm 2 - Treatment Group Prosthetists, Pre and Post Modifications; Arm 2 - Control Group Prosthetists, Pre and Post Modifications: Participant's in Arm 2 had their prosthetists recruited as well. Prosthetists for participants in both control and treatment groups were surveyed regarding modifications to their patient's socket. Prosthetists for participants in Arm 2 were also given pre-modification bioImpedance data as a supplement to their socket modification process and were surveyed regarding this data as well.
- Total: Total of all reporting groups
Arm/Group | Arm 1 - Pre and Post Modification Observation, No Intervention | Arm 2 - Treatment Group, Pre and Post Modification | Arm 2 - Control Group, Pre and Post Modification | Arm 2 - Treatment Group Prosthetists, Pre and Post Modifications | Arm 2 - Control Group Prosthetists, Pre and Post Modifications | Total
Number analyzed (Participants) | 19 | 16 | 16 | 8 | 9 | 68
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 17 | 11 | 12 | 8 | 9 | 57
  >=65 years | 2 | 5 | 4 | 0 | 0 | 11
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 2 | 1 | 2 | 11
  Male | 16 | 13 | 14 | 7 | 7 | 57
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 0 | 0 | 1
  Not Hispanic or Latino | 19 | 15 | 16 | 8 | 9 | 67
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 0 | 0 | 0 | 0 | 3
  Asian | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 0 | 0 | 1
  Black or African American | 1 | 1 | 2 | 0 | 0 | 4
  White | 15 | 13 | 13 | 8 | 9 | 58
  More than one race | 0 | 1 | 0 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 1 | 0 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 19 | 16 | 16 | 8 | 9 | 68

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Significant Increases in Socket Comfort Score (SCS)
Description: Participants are asked to quantify the overall comfort of their prosthesis by giving it a score between 0 and 10 with 0 as the least comfortable possible and 10 being the most comfortable possible. SCS scores were acquired both pre and post making modifications to the participant's prosthesis. For analysis purposes, the number of participants that had a significant positive change are counted for this outcome. Participants that had little to no change (a score difference <2) in SCS or had a negative change in SCS score were not counted.
Time Frame: Baseline taken pre-modification, with a final score taken post-modification. The minimum time between scores was 3 weeks.
Population: Primary outcome measures from each group were collected pre and post modifications to their prosthesis. The experimental arm involved sharing bioimpedance data with the participants' prosthetist.
Measure: Number; unit: participants
Groups:
- Arm 2 - Treatment: Conclusions drawn from data gathered in Arm 1 will be given to the participant's prosthetist, along with their bioimpedance data from Arm 2, to inform the practitioner's decision on when a modification to the socket is warranted. The results will be compared to those of Arm 3.
  Bioimpedance monitor: Participant in aim 1 will be monitored using the bioimpedance monitor. Data obtained from the arm 1 cohort will be used to inform socket modifications made for arm 2 cohort.
Arm/Group | Arm 1 | Arm 2 - Treatment | Arm 3 - Control
Number analyzed (Participants) | 14 | 10 | 11
participants | 5 | 6 | 4

2. Secondary Outcome: Number of Participants With Net-Positive Increase in Prosthesis Satisfaction, Measured by the Patient's Overall Satisfaction With Their Entire Prosthesis
Description: Participants are asked to indicate their overall satisfaction with their prosthesis by drawing a line on a continuous scale running from extremely unhappy to extremely happy (0 to 100). For analysis purposes, the number of participants that had a net positive change are counted for this outcome. Participants that had a net negative or no change were not counted.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 - Pre and Post Modification Observation, No Intervention | Arm 2 - Treatment Group, Pre and Post Modification | Arm 2 - Control Group, Pre and Post Modification
Number analyzed (Participants) | 14 | 10 | 11
Participants | 8 | 6 | 6

3. Secondary Outcome: Number of Participants With Net-Positive Change in Ambulation Score
Description: Participants are asked to indicate their overall ability to walk with their prosthesis by drawing a line on a continuous scale running from "Cannot Walk at All" to "No Problem Walking" (0 to 100, respectively). They are also asked questions related to ambulation ability in unique circumstances, such as walking in close spaces, up and down stairs, up and down hills, on streets, on sidewalks, and on slippery surfaces. For analysis purposes, the number of participants that had a net positive change are counted for this outcome. Participants that had a net negative or no change were not counted.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 - Pre and Post Modification Observation, No Intervention | Arm 2 - Treatment Group, Pre and Post Modification | Arm 2 - Control Group, Pre and Post Modification
Number analyzed (Participants) | 14 | 10 | 11
Participants | 11 | 8 | 8

4. Secondary Outcome: Number of Participants With Net-Positive Change in Residual Limb Health Score
Description: Participants are asked to indicate how much their residual limb sweats, smells, swells, develops rashes, develops ingrown hairs, and develops blisters, while wearing their prosthesis.They indicate this by drawing a line on a continuous scale running from "Extreme Amount" to "Not At All" (0 to 100, respectively). For analysis purposes, the number of participants that had a net positive change are counted for this outcome. Participants that had a net negative or no change were not counted.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 - Pre and Post Modification Observation, No Intervention | Arm 2 - Treatment Group, Pre and Post Modification | Arm 2 - Control Group, Pre and Post Modification
Number analyzed (Participants) | 14 | 10 | 11
Participants | 10 | 3 | 6

5. Secondary Outcome: Number of Participants With Net-Positive Change in Prosthesis Utility Score
Description: Participants are asked to indicate various features related to the utility of their prosthesis by drawing a line on a continuous scale that ranges from "Terrible" to "Excellent" (0 to 100, respectively). Features include prosthesis fit, weight, comfort while standing, comfort while sitting, balance, effort, feel, and donning. For analysis purposes, the number of participants that had a net positive change are counted for this outcome. Participants that had a net negative or no change were not counted.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 - Pre and Post Modification Observation, No Intervention | Arm 2 - Treatment Group, Pre and Post Modification | Arm 2 - Control Group, Pre and Post Modification
Number analyzed (Participants) | 14 | 10 | 11
Participants | 11 | 9 | 9

6. Secondary Outcome: Number of Participants With Net-Positive Change in Prosthesis Well Being Score
Description: Prosthesis users indicate their well being since their amputation and also rank their overall quality of life by marking a line on a scale ranging from "worst possible life" to "best possible life" (0 to 100, respectively). Participants who showed a positive net increase in this category were counted for each aim.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 - Pre and Post Modification Observation, No Intervention | Arm 2 - Treatment Group, Pre and Post Modification | Arm 2 - Control Group, Pre and Post Modification
Number analyzed (Participants) | 14 | 10 | 11
Participants | 8 | 7 | 6

7. Secondary Outcome: Prosthetist Communication Assessment Score, Measured by the Communication Efficacy Between the Prosthetist and Their Patient
Description: Participants' prosthetists are asked to rate their ability to communicate the need for sock or behavioral changes to their patients participating in the study. They will indicate the score using a scale from 0 to 10 with 10 being the best possible communication and 0 being the worst possible communication.
Time Frame: Baseline, prior to socket modification
Population: Only participants that completed surveys both pre and post modifications to their patient's sockets were included in this analysis.
Measure: Mean (Full Range); unit: score on a scale
Groups:
- Arm 2 - Treatment Group Prosthetists, Pre Modifications; Arm 2 - Control Group Prosthetists, Pre-Modifications: Participant's in Arm 2 had their prosthetists recruited as well. Prosthetists for participants in both control and treatment groups were surveyed regarding modifications to their patient's socket. Prosthetists for participants in Arm 2 were also given pre-modification bioImpedance data as a supplement to their socket modification process and were surveyed regarding this data as well.
Arm/Group | Arm 2 - Treatment Group Prosthetists, Pre Modifications | Arm 2 - Control Group Prosthetists, Pre-Modifications
Number analyzed (Participants) | 8 | 9
score on a scale | 9 [8 to 10] | 8.8 [7 to 10]

8. Secondary Outcome: Types of Socket Modifications Implemented Per Group
Description: Participants' prosthetists are asked the type of socket modification(s) that they implemented in free response format. Responses were simplified into 5 categories related to common modification changes. The most common themes were: fabrication of a new socket, addition of socket pads or an insert, creating socket reliefs, changing socket suspension, and other. Changes that fell under the "other" category were not necessarily related to changes in socket shape, such as changes in overall prosthesis alignment, prosthesis foot, fabrication materials, etc.
Time Frame: Baseline, prior to socket modification
Population: Only participants who completed the survey and whose patients completed pre and post-modification testing were included in this analysis. Prosthetists' responses from both the control and treatment groups are counted for this metric. Some prosthetists had more than one participant in the study which may impact total counts for this metric.
Measure: Count of Participants; unit: Participants
Groups:
- Arm 2 - Treatment Group, Pre and Post Modification: Participants' socket modifications were based only on their prosthetists. Prosthetists for this group did not receive any bioimpedance data to inform their decisions.
- Arm 2 - Control Group, Pre and Post Modification: Participants' socket modifications were based on their prosthetists after said prosthetists received bioimpedance data.
Arm/Group | Arm 2 - Treatment Group, Pre and Post Modification | Arm 2 - Control Group, Pre and Post Modification
Number analyzed (Participants) | 10 | 11
Participants
  New Socket | 9 | 11
  Socket pad/insert | 1 | 3
  socket relief | 0 | 1
  Suspension change | 1 | 1
  Other | 6 | 1

9. Secondary Outcome: Effect of Socket Modification, Measured by the Impact of the Physical Modification Made to the Prosthesis to Socket Fit
Description: Participants' prosthetists from both groups were asked to rate the effectiveness of the modification(s) that they implemented on a scale of 0 to 10 in which 10 is "Excellent" and 0 is "Terrible".
Time Frame: Post modification, minimum 4 weeks after patient started study
Population: Only participants who completed the survey and whose patients completed pre and post modification treatment group testing were included in this analysis.
Measure: Mean (Full Range); unit: score on a scale
Groups:
- Arm 2 - Treatment Group Prosthetists, Post Modifications; Arm 2 - Control Group Prosthetists, Post-Modifications: Participant's in Arm 2 had their prosthetists recruited as well. Prosthetists for participants in both control and treatment groups were surveyed regarding modifications to their patient's socket. Prosthetists for participants in Arm 2 were also given pre-modification bioImpedance data as a supplement to their socket modification process and were surveyed regarding this data as well.
Arm/Group | Arm 2 - Treatment Group Prosthetists, Post Modifications | Arm 2 - Control Group Prosthetists, Post-Modifications
Number analyzed (Participants) | 8 | 9
score on a scale | 8.3 [3 to 10] | 8.6 [5 to 10]

10. Secondary Outcome: Strategies Recommended to Minimize Limb Fluid Volume Loss
Description: Participants' prosthetists are asked what changes to the participant's volume management strategy they recommended in free-response format. The following common themes were pulled from their responses: new sock regimen, periodic doffing, new activity regimen, new self-care regimen, other, and none. A count for how many prosthetists mentioned the same theme was tabulated.
Time Frame: Post modification, minimum 4 weeks after patient started study
Population: Only participants who completed the survey and whose patients completed pre and post modification testing were included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 2 - Treatment Group Prosthetists, Post Modifications | Arm 2 - Control Group Prosthetists, Post-Modifications
Number analyzed (Participants) | 8 | 9
Participants
  New Sock Regimen | 2 | 3
  Periodic Doffing | 3 | 1
  Activity Regimen | 0 | 0
  Self-Care Regimen | 0 | 0
  Other | 0 | 0
  None | 2 | 2

11. Secondary Outcome: Effect of Volume Management Strategy, Measured by the Impact of the Changes in Volume Management to Socket Fit
Description: Participants' prosthetists are asked to rate the effectiveness of the strategies that they recommended on a scale of 0 to 10 in which 10 is "Excellent" and 0 is "Terrible".
Time Frame: Post modification, minimum 4 weeks after patient started study
Population: Only participants who completed the survey and whose patients completed pre and post modification testing were included in this analysis. Note: two control group prosthetists did not provide an answer for this portion of the survey.
Measure: Mean (Full Range); unit: score on a scale
Groups:
- Arm 2 - Control Group Prosthetists, Post Modifications: Participant's in Arm 2 had their prosthetists recruited as well. Prosthetists for participants in both control and treatment groups were surveyed regarding modifications to their patient's socket. Prosthetists for participants in Arm 2 were also given pre-modification bioImpedance data as a supplement to their socket modification process and were surveyed regarding this data as well.
Arm/Group | Arm 2 - Treatment Group Prosthetists, Post Modifications | Arm 2 - Control Group Prosthetists, Post Modifications
Number analyzed (Participants) | 8 | 7
score on a scale | 6.3 [0 to 8] | 6.7 [5 to 9]

12. Secondary Outcome: Modification/Strategy Satisfaction, Measured by Overall Satisfaction of All Methods Employed
Description: Prosthetists are asked to rate their overall satisfaction with the socket modification and/or volume management change that was used for each participant by indicating a score from 0 to 10 with 10 being "Extremely Satisfied" and 0 being "Not Satisfied".
Time Frame: Post modification, minimum 4 weeks after patient started study
Population: as for outcome 10
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Arm 2 - Treatment Group Prosthetists, Post Modifications | Arm 2 - Control Group Prosthetists, Post-Modifications
Number analyzed (Participants) | 8 | 9
score on a scale | 8.4 [7 to 10] | 7.9 [5 to 10]

13. Secondary Outcome: Prosthetist Impression of Bioimpedance Results, Measured by General Feedback From Clinicians on the Bioimpedance Data They Are Given
Description: Prosthetists are asked to describe their impression of the bioimpedance results in a free response format. Common themes were gathered from responses and a count for each was tabulated based on gathered responses.
Time Frame: Post modification, minimum 4 weeks after patient started study
Population: Only participants who completed the survey and whose patients completed pre and post modification testing in the "Treatment" group were included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 2 - Treatment Group Prosthetists, Post Modifications
Number analyzed (Participants) | 8
Participants
  Found results helpful/interesting | 4
  Results aligned with physiological expectations | 3
  Results did not align with physiological expectations | 2
  Highlighted detail of results | 4

14. Secondary Outcome: Prosthetist Use of Bioimpedance Results, Measured by General Feedback on How the Clinicians Use the Bioimpedance Data They Are Given
Description: Prosthetists are asked to describe, in free response format how they used the bioimpedance results to inform their clinical practice. Common themes were gathered from responses and a count for each was tabulated based on gathered responses.
Time Frame: Post modification, minimum 4 weeks after patient started study
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 2 - Treatment Group Prosthetists, Post Modifications
Number analyzed (Participants) | 8
Participants
  To discuss daily activity patterns with patient | 2
  To communicate socket management topics with patient | 3
  To communicate physiological issues with patient | 3
  To inform socket modifications | 2
  Unsure/Did Not Use | 1

15. Secondary Outcome: Bioimpedance Usefulness for Socket Design, Measured by General Feedback on How Useful Bioimpedance is for Informing Decisions on Socket Modifications
Description: Participants' prosthetists are asked to rate the effectiveness of the strategies that they recommended on a scale of 0 to 10 in which 10 is "Very Useful" and 0 is "Not Useful".
Time Frame: Post modification, minimum 4 weeks after patient started study
Population: as for outcome 13
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Arm 2 - Treatment Group Prosthetists, Post Modifications
Number analyzed (Participants) | 8
score on a scale | 6.9 [0 to 10]

16. Secondary Outcome: Bioimpedance for Volume Management, Measured by General Feedback on How Useful Bioimpedance is for Informing Decisions on Socket Modifications
Description: Prosthetists are asked to rate the utility of bioimpedance results in recommending volume management strategies to their patients. The rating scale is 0 to 10 with 10 being "Very Useful" and 0 being "Not Useful".
Time Frame: Post modification, minimum 4 weeks after patient started study
Population: Only participants who completed the survey and whose patients completed pre and post-modification testing in the "Treatment" group were included in this analysis.
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Arm 2 - Treatment Group Prosthetists, Post Modifications
Number analyzed (Participants) | 8
score on a scale | 8.3 [5 to 10]

17. Secondary Outcome: Continuing Use of Bioimpedance Results, Measured by How Likely Clinicians Will be to Use Bioimpedance Data in the Future
Description: Prosthetists are asked to indicate how likely they are to request bioimpedance data for their other patients by selecting a score from 0 to 10 with 10 with being "Very Likely" and 0 being "Not Likely at All".
Time Frame: Post modification, minimum 4 weeks after patient started study
Population: as for outcome 13
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Arm 2 - Treatment Group Prosthetists, Post Modifications
Number analyzed (Participants) | 8
score on a scale | 8.5 [6 to 10]

18. Secondary Outcome: Impact of Bioimpedance, Measured by How Bioimpedance Data Changed the Way Prosthetists Approach Problem Issues of Socket Fit
Description: Prosthetists are asked to quantify the impact that the bioimpedance had on the manner in which they approached the issue by rating the impact from 0 to 10 with 10 being "Very Impactful" and 0 being "No Impact".
Time Frame: Post modification, minimum 4 weeks after patient started study
Population: as for outcome 13
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Arm 2 - Treatment Group Prosthetists, Post Modifications
Number analyzed (Participants) | 8
score on a scale | 5.9 [0 to 10]

19. Secondary Outcome: Most Useful Bioimpedance Data, Measured by Which Element of the Bioimpedance Data is Most Useful to Clinicians
Description: Prosthetists are asked to select from a list which bioimpedance data was most useful to them. The list items are: magnitude of fluid volume change over the whole day, fluid volume change by regions of the limb, fluid volume change from different activities, rate of fluid volume change over the whole day, and rate of fluid volume change over specific activity intervals
Time Frame: Post modification, minimum 4 weeks after patient started study
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 2 - Treatment Group Prosthetists, Post Modifications
Number analyzed (Participants) | 8
Participants
  magnitude of fluid volume change over the whole day: Identified as useful | 4
  magnitude of fluid volume change over the whole day: Did not identify as useful | 4
  fluid volume change by regions of the limb: Identified as useful | 3
  fluid volume change by regions of the limb: Did not identify as useful | 5
  fluid volume change from different activities: Identified as useful | 6
  fluid volume change from different activities: Did not identify as useful | 2
  rate of fluid volume change over the whole day: Identified as useful | 4
  rate of fluid volume change over the whole day: Did not identify as useful | 4
  rate of fluid volume change over specific activity intervals: Identified as useful | 4
  rate of fluid volume change over specific activity intervals: Did not identify as useful | 4
  Other (pressure mapping based on limb volume): Identified as useful | 1
  Other (pressure mapping based on limb volume): Did not identify as useful | 7

20. Secondary Outcome: Bioimpedance and Communication Measured by General Feedback on Whether Prosthetist-patient Communication is Improved Through Use of Bioimpedance Data
Description: Prosthetists are asked to indicate the degree to which their use bioimpedance results improved the communication between them and their patients. They indicate this by selecting a value from 0 to 10 with 10 being "Highly Impactful" and 0 being "No Impact".
Time Frame: Post modification, minimum 4 weeks after patient started study
Population: as for outcome 13
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Arm 2 - Treatment Group Prosthetists, Post Modifications
Number analyzed (Participants) | 8
score on a scale | 8.1 [6 to 10]

21. Secondary Outcome: Outcome Enhancement, Measured by the Degree to Which Outcomes Are Improved Using Bioimpedance Data
Description: Prosthetists are asked to indicated the degree to which clinical outcomes were enhanced by the use of bioimpedance results. They indicate this by selecting a value from 0 to 10 with 10 being "Positive Impact" and 0 being "Negative Impact".
Time Frame: Post modification, minimum 4 weeks after patient started study
Population: as for outcome 13
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Arm 2 - Treatment Group Prosthetists, Post Modifications
Number analyzed (Participants) | 8
score on a scale | 6.6 [2 to 9]

ADVERSE EVENTS:
Time Frame: through study completion, 4 years
Description: Adverse Events were monitored/assessed, but none observed
Arm/Group | Arm 1 - Pre and Post Modification Observation, No Intervention | Arm 2 - Treatment Group, Pre and Post Modification | Arm 2 - Control Group, Pre and Post Modification | Arm 2 - Treatment Group Prosthetists, Pre and Post Modifications | Arm 2 - Control Group Prosthetists, Pre and Post Modifications
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/16 | 0/16 | 0/8 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/16 | 0/16 | 0/8 | 0/9
Other Adverse Events (participants affected / at risk) | 0/17 | 0/16 | 0/16 | 0/8 | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-04-27): https://cdn.clinicaltrials.gov/large-docs/56/NCT03164356/Prot_SAP_001.pdf